CLINICAL TRIAL: NCT02895620
Title: Evaluation of the Effect of a Complex Inflammatory Milieu Induced by BCG Treatment in Urines of Patients With Non-muscle-invasive Bladder Cancer on the Xpert® Bladder Cancer Assay
Brief Title: Effect on Xpert® Bladder Test of Urines Inflammatory Milieu Induced by BCG Treatment of Patients With NMIBC
Acronym: CEPHEID
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institut Claudius Regaud (Other)
Collaborators: Cepheid (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 16HLURO01
Record Dates: First submitted 2016-09-06; First posted 2016-09-09 (Estimated); Last update posted 2016-09-09 (Estimated); Status verified 2016-09

CONDITIONS: Non Muscle Invasive Bladder Cancer; Treatment by BCG
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NMIBC patients Xpert bladder test (Other): Xpert bladder test of urine of patients with NMIBC treated with BCG therapy
  Interventions: Biological: Xpert bladder Test

INTERVENTIONS:
Biological: Xpert bladder Test — Xpert test positive or negative on urine samples of NMIBC patients treated by BCG

SUMMARY:
Intravesical BCG immunotherapy is used after transurethral resection (TUR) for the prevention of recurrence of NMIBC. BCG treatment is usually started a few weeks after TUR and is given once a week for 6 weeks. It stimulates immune responses that can destroy bladder cancer cells (acute and chronic induced inflammations) and as a consequence causes side effects. The investigators postulate that Xpert® test might be used to demonstrate the presence of residual (after TURB) or recurrent (during adjuvant treatment) disease at the time of intravesical treatment, which could be of very significant impact in the management of this complex situation.Urines of BCG treated patients are rich in immune system elements (cytokines, lymphocytes,…), this complex inflammatory milieu of urines may interfere with urinary biomarkers. This study will allow assessing the effect of the complex inflammatory milieu induced by BCG treatment in urines of patients with NMIBC on the Xpert® Bladder cancer assay.

DETAILED DESCRIPTION:
1. Qualification of Xpert® Testing:

   Three 50 mL fresh urine samples will be collected in sterile containers according to Cepheid instructions of use:
   * the "baseline sample" before the first BCG instillation,
   * the "study sample" taken during the initiation course of treatment instillations, preferably at the 4th or 5th instillation of BCG therapy,
   * the "follow-up sample" at the time of the first follow-up cystoscopy, approximately 3 months after the last BCG instillation of the initiation course.

   Xpert® test results will be qualified as positive or negative, according to Cepheid instructions for use.

   Samples tested positive at baseline will not be included in the analysis and the patient's participation in the study will be discontinued.

   Samples obtained in patients with no recurrence at follow-up cystoscopy after the initiation course will be considered for analysis.
2. Threshold of detection of theXpert® Bladder test:

   * One urine sample of a patient tumor free (negative Xpert test) under BCG treatment will be spiked into 3 log dilutions of the 2 distinct tumor cell lines SW780 and BE(2)-C (100, 1000, and 10000 cells per ml).
   * A mix of fresh and frozen cells from en bloc harvested tumors from distinct donors will be tested at the set concentration in BCG urines from distinct patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with high-risk transitional cell carcinoma of the bladder, according to the EAU guidelines/EORTC risk stratification, who are offered adjuvant BCG instillations.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Rate of negative Xpert tests results during the initiation course in patients with no recurrence at first follow-up cystoscopy | 12 months

SECONDARY OUTCOMES:
rate of Xpert tests found positive in samples with predefined tumour cell concentrations ( limit of detection) in inflammatory milieu of urines induced by the BCG treatment in patients with bladder cancer | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institut claudius regaud IUCT ONCOPOLE, Toulouse, France

IPD SHARING:
Plan to Share IPD: No